CLINICAL TRIAL: NCT02098733
Title: Pioglitazone/Glimepiride (Sonias) Combination Tablets Special Drug Use Surveillance Survey on Long-term Use for in Type 2 Diabetes Mellitus
Brief Title: Long-term Use of Sonias Combination Tablets in Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 097-011; JapicCTI-142438 (Registry Identifier: Japic CTI); JapicCTI-R150734 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
Keywords: Pharmacological therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; glimepiride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pioglitazone/glimepiride: Pioglitazone/glimepiride 15 mg/1 mg or 30 mg/3 mg, orally once daily before or after breakfast
  Interventions: Drug: Pioglitazone/glimepiride

INTERVENTIONS:
Drug: Pioglitazone/glimepiride — Pioglitazone/glimepiride combination tablets
  Other Names: Sonias combination tablets

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term use of Sonias Combination Tablets in patients with type 2 diabetes mellitus in the routine clinical setting.

DETAILED DESCRIPTION:
This a special drug use surveillance on long-term use of pioglitazone/glimepiride combination tablets (Sonias Combination Tablets) designed to investigate the frequency of adverse drug reactions in patients with type 2 diabetes mellitus in the routine clinical setting.

The usual adult dosage is one tablet of Sonias administered orally once daily before or after breakfast (15 mg/1 mg or 30 mg/3 mg of pioglitazone/glimepiride).

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus for whom a physician has concluded that combination therapy with pioglitazone hydrochloride and glimepiride is appropriate and for whom long-term treatment with Sonias Combination Tablets is considered necessary

Exclusion Criteria:

* (1) Patients with cardiac failure or a history of cardiac failure (2) Patients with serious hepatic or renal impairment (3) Patients with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus (4) Patients with severe infection, severe trauma, or pre- and post-operative patients (5) Patients with gastrointestinal disorders such as diarrhea and vomiting (6) Pregnant or potentially pregnant women (7) Patients with a history of hypersensitivity to the ingredients in Sonias Combination Tablets or sulfonamides

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1168 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 182 investigative sites in Japan from 15 June 2011 to 31 May 2014.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus for whom therapy with pioglitazone combined with glimepiride is suitable and long-term treatment is considered necessary were enrolled in one treatment group to receive pioglitazone/glimepiride 15 mg/1 mg or 30 mg/3 mg, orally once daily before or after breakfast.
Period: Overall Study
Arm/Group | Pioglitazone/Glimepiride
Started | 1168
Completed | 1158
Not Completed | 10
Not completed — Data Not Available | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants with available data.
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 1158
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (12.14)
Age, Customized [Number; unit: participants]
  <65 years | 539
  ≥65 years | 619
Age, Customized [Number; unit: participants]
  <65 years | 539
  ≥65 to <74 years | 354
  ≥75 years | 265
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 439
  Male | 719
Pregnancy Status <Females> [Number; unit: participants] — Female participants only (n=439)
  participants
    Not pregnant | 439
    Pregnant | 0
Weight [Mean (Standard Deviation); unit: kg] | 67.86 (14.281)
Weight Categorical [Number; unit: participants]
  <40 kg | 7
  ≥40 to <50 kg | 74
  ≥50 to <60 kg | 223
  ≥60 to <70 kg | 327
  ≥70 kg | 427
  Unmeasured | 100
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data was available for 1011 participants.
  kg/m^2 | 26.19 (4.401)
BMI Categorical [Number; unit: participants]
  <18.5 kg/m^2 | 12
  ≥18.5 to <25 kg/m^2 | 422
  ≥25 to <30 kg/m^2 | 412
  ≥30 kg/m^2 | 165
  Unknown | 147
Duration of Type 2 Diabetes [Mean (Standard Deviation); unit: years] — Duration of type 2 diabetes data was available for 788 participants.
  years | 9.12 (8.188)
Duration of Type 2 Diabetes, Categorical [Number; unit: participants]
  <2 years | 92
  ≥2 to <5 years | 160
  ≥5 to <10 years | 262
  ≥10 years | 274
  Unknown | 370
Healthcare Category [Number; unit: participants]
  Outpatient | 1155
  Inpatient | 3
History of Allergies [Number; unit: participants]
  No | 959
  Yes | 81
  Unknown | 118
Presence of Complications [Number; unit: participants]
  No | 108
  Yes | 1050
Breakdown of Complications [Number; unit: participants] — Participants may be accounted for in more than 1 category.
  participants
    Microangiopathy | 227
    Diabetic nephropathy | 144
    Diabetic retinopathy | 71
    Diabetic neuropathy | 88
    Hypertension | 723
    Dyslipidaemia | 787
    Hyperuricaemia | 95
    Liver disease | 154
    Renal disease | 159
    Heart disease | 134
    Cerebrovascular disease | 76
    Malignant tumor | 10
    Other | 19
Presence of Medical History [Number; unit: participants]
  No | 897
  Yes | 157
  Unknown | 104
Alcohol History (Drinking Alcohol-Containing Beverages Most Days) [Number; unit: participants]
  Yes | 596
  No | 375
  Unknown | 187
Smoking Classification [Number; unit: participants]
  Never Smoked | 516
  Current Smoker | 191
  Ex-smoker | 228
  Unknown | 223
Compliance Rate with the Diet Regimen (At the Start of Treatment) [Number; unit: participants]
  ≥ 90% | 285
  ≥ 70% | 371
  ≥ 50% | 286
  < 50% | 91
  Undone or compliance status is unknown | 125
Compliance rate with the Exercise Regimen (At the Start of Treatment) [Number; unit: participants]
  ≥ 90% | 219
  ≥ 70% | 279
  ≥ 50% | 348
  < 50% | 147
  Undone or compliance status is unknown | 165
Timing of Initiation of Pioglitazone Before the Start of Study Treatment [Number; unit: participants] — Data is only available for participants who were administered pioglitazone alone prior to beginning study treatment (n=189).
  participants
    ≥ 3 months | 104
    < 3 months | 17
    Unknown | 68
Timing of Initiation of Glimepiride Before the Start of Study Treatment [Number; unit: participants] — Data is only available for participants who were administered glimepiride alone prior to beginning study treatment (n=338).
  participants
    ≥ 3 months | 223
    < 3 months | 42
    Unknown | 73
Timing of Initiation of Pioglitazone and Glimepiride Before the Start of Study Treatment [Number; unit: participants] — Data is only available for participants who were administered both pioglitazone and glimepiride prior to beginning study treatment (n=558).
  participants
    ≥ 3 months | 347
    Other | 60
    Unknown | 151
Glycosylated Haemoglobin (HbA1c) at the Start of Study Treatment [Number; unit: participants]
  < 6.0% | 35
  ≥ 6.0% to < 7.0% | 274
  ≥ 7.0% to < 8.0% | 427
  ≥ 8.0% | 355
  Unknown | 67
HbA1c at the Start of Study Treatment [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] — HbA1c data was available for 1091 participants.
  percentage of glycosylated haemoglobin | 7.71 (1.313)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: Adverse events are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: For 12 months
Population: All enrolled participants with available data.
Measure: Number; unit: participants
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 1158
participants
  Hypoglycaemia | 13
  Dizziness | 4
  Dysgeusia | 1
  Headache | 1
  Hypoaesthesia | 1
  Cardiac failure | 2
  Cardiac failure congestive | 1
  Pleural effusion | 1
  Eructation | 1
  Nausea | 1
  Cholelithiasis | 1
  Drug eruption | 1
  Pruritus | 2
  Swelling face | 1
  Urticaria | 1
  Face oedema | 1
  Feeling abnormal | 1
  Hunger | 2
  Oedema | 7
  Oedema peripheral | 4
  Sudden death | 1
  Blood creatine phosphokinase increased | 1
  Alanine aminotransferase increased | 1
  Blood triglycerides increased | 1
  Blood glucose decreased | 1
  Weight increased | 8

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Tabulated the changes from baseline in glycosylated hemoglobin (HbA1c) values at each test time point (test value at each test time point after baseline - test value at baseline). A negative change from Baseline indicates improvement.
Time Frame: Baseline, and Months 3, 6, 9, 12 and at Final Assessment
Population: All enrolled participants with data available.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 1059
percentage of glycosylated haemoglobin
  Month 3 (n=1016) | -0.45 (0.936)
  Month 6 (n=893) | -0.55 (1.144)
  Month 9 (n=831) | -0.56 (1.107)
  Month 12 (n=462) | -0.57 (1.196)
  Final Assessment (n=1,054) | -0.57 (1.152)

3. Secondary Outcome: Glycosylated Hemoglobin (HbA1c)
Description: Tabulated glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at each test time point or final visit relative to baseline.
Time Frame: Baseline, and Months 3, 6, 9, 12 and at Final Assessment
Population: All enrolled participants with data available.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 1059
percentage of glycosylated haemoglobin
  At the start of treatment (n=1054) | 7.70 (1.302)
  Month 3 (n=1016) | 7.25 (1.102)
  Month 6 (n=893) | 7.14 (1.059)
  Month 9 (n=831) | 7.08 (0.995)
  Month 12 (n=462) | 7.12 (1.077)
  Final Assessment (n=1054) | 7.13 (1.100)

4. Secondary Outcome: Change From Baseline in Fasting Blood Glucose Level
Description: Tabulated the changes from baseline in fasting blood glucose level at each test time point (test value at each test time point after baseline - test value at baseline). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3, 6, 9, 12 and at Final Assessment
Population: All enrolled participants with data available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 1059
mg/dL
  Month 3 (n=331) | -16.7 (44.39)
  Month 6 (n=287) | -14.3 (48.17)
  Month 9 (n=273) | -15.7 (45.94)
  Month 12 (n=462) | -12.5 (45.50)
  Final Assessment (n=369) | -16.4 (47.41)

5. Secondary Outcome: Fasting Blood Glucose Level
Description: Tabulated fasting blood glucose level from baseline at each test time point.
Time Frame: Baseline, Months 3, 6, 9, 12 and at Final Assessment
Population: All enrolled participants with data available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 1059
mg/dL
  At the start of treatment (n=369) | 147.2 (51.87)
  Month 3 (n=331) | 130.2 (43.18)
  Month 6 (n=287) | 131.7 (41.09)
  Month 9 (n=273) | 129.2 (36.71)
  Month 12 (n=462) | 126.8 (42.01)
  Final Assessment (n=369) | 130.9 (46.82)

6. Secondary Outcome: Change From Baseline in Fasting Insulin Level
Description: Tabulated the changes from baseline at each test time point (test value at each test time point after baseline - test value at baseline). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Months 3, 6, 9, 12 and at Final Assessment
Population: All enrolled participants with data available.
Measure: Mean (Standard Deviation); unit: μU/dL
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 1059
μU/dL
  Month 3 (n=39) | -0.24 (1.376)
  Month 6 (n=32) | 0.02 (1.163)
  Month 9 (n=30) | -0.60 (2.121)
  Month 12 (n=18) | 0.58 (2.582)
  Final Assessment (n=46) | -0.01 (2.397)

7. Secondary Outcome: Fasting Insulin Level
Description: Tabulated fasting insulin level at each test time point.
Time Frame: Baseline, Months 3, 6, 9, 12 and at Final Assessment
Population: All enrolled participants with data available.
Measure: Mean (Standard Deviation); unit: μU/dL
Arm/Group | Pioglitazone/Glimepiride
Number analyzed (Participants) | 1059
μU/dL
  At the start of treatment (n=46) | 5.78 (2.880)
  Month 3 (n=39) | 5.38 (2.885)
  Month 6 (n=32) | 5.48 (2.964)
  Month 9 (n=30) | 5.40 (2.642)
  Month 12 (n=18) | 6.57 (3.789)
  Final Assessment (n=46) | 5.77 (3.238)

ADVERSE EVENTS:
Time Frame: For 12 months
Description: At each visit the investigator documented any occurrence of adverse events and abnormal laboratory findings. Any event reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Pioglitazone/Glimepiride
Serious Adverse Events (participants affected / at risk) | 23/1158
Other Adverse Events (participants affected / at risk) | 0/1158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone/Glimepiride (N=1158)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Death (General disorders) | 1
Drowning (General disorders) | 1
Face oedema (General disorders) | 1
Oedema (General disorders) | 1
Sudden death (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.